CLINICAL TRIAL: NCT01512277
Title: Phase 1 Study Evaluating Safety and Immunological Criteria of Efficacy of the Recombinant Vaccine Candidate Bilhvax Against Schistosomiasis
Brief Title: Clinical Trial of Bilhvax,a Vaccine Candidate Against Schistosomiasis
Acronym: Bilhvax1a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP97/104; 98002 (Other: Sponsor); 980056 (Other: DGS)
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Schistosomiasis; Bilharziasis; Urinary Schistosomiasis
Keywords: vaccines; safety; drug tolerance; immunogenic protein; antibody response; cytokine
MeSH Terms: conditions — Schistosomiasis; Schistosomiasis haematobia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 administrations of 100 µg of rSh28GST (Experimental): Adult volunteers (n=8) receive 100μg of rSh28GST together with aluminium hydroxide (Alum) as adjuvant at D0, D28, and D150.
  Interventions: Biological: rSh28GST
- 2 administrations of 300 µg of rSh28GST (Experimental): Adult volunteers (n=8) receive 300μg of rSh28GST together with aluminium hydroxide (Alum) as adjuvant at D0 and D28.
  Interventions: Biological: rSh28GST
- Placebo (Placebo Comparator): Adult volunteers (n=8) receive aluminium hydroxide (Alum) alone at D0 and D28.
  Interventions: Biological: rSh28GST

INTERVENTIONS:
Biological: rSh28GST — subcutaneous route at Day 0, Day 28, and Day 150 for the third administration of 100µg for Arm 1
  Other Names: Bilhvax

SUMMARY:
The purpose of this clinical study is to evaluate safety and immunogenicity in adult healthy volunteers of the vaccine candidate against schistosomiasis named Bilhvax.

DETAILED DESCRIPTION:
The development of an efficient vaccine against human schistosomiasis represents a major challenge for the improvement of health in many developing countries.

Schistosomiasis affects millions people in numerous countries and hampers economical development of tropical areas.

Although progress has been made for the limitation of the disease severity by chemotherapy, continuous re-infection and risks of drug resistance point to the necessary development of alternative strategies.

It is widely agreed that immunological prevention of chronic parasitic infections will be extremely difficult to achieve. Conversely in some major helminth infections like schistosomiasis, where parasite eggs laying in the tissues is the exclusive cause of pathology and the elimination of eggs in nature is the source of transmission, inhibition of parasite fecundity might represent for the future a novel way to prevent the deleterious effects of these chronic infections in man.

The concept to target by vaccination the cause of the pathology rather than the parasite itself would provide a potent tool to control a major chronic infection.

After years of basic studies on effector and regulatory mechanisms of immune response against schistosomiasis it has been identify a schistosome molecule named glutathione S-transferase 28 kDa (28GST) presenting a potential as vaccine candidate.

This 28GST have been cloned and named Bilhvax. It has been shown that immunization with such schistosome GST would dramatically decrease female worm fecundity and egg viability in various hosts. It was demonstrated that these anti-fecundity effects are associated with the production of antibodies neutralizing the GST enzymatic activities obtained through a Th2-type immune response. This correlation between anti-fecundity effects and inhibition-mediated antibodies demonstrated in several animal models was re-enforced by epidemiological studies showing that such acquired antibodies produced during infection could be detected in adult individuals naturally resistant to the re-infection.

The present phase 1 clinical trial is conducted in healthy Caucasian volunteers to evaluate as primary endpoint the safety of the recombinant Sh28GST (rSh28GST) in Alum (named Bilhvax), a vaccine candidate against human urinary schistosomiasis. The secondary endpoint is to evaluate immunogenicity of Bilhvax, to determine the profile of the immune response, and to estimate the neutralizing capacity of the antibodies against the rSh28GST enzymatic activity.

The recombinant S. haematobium 28GST expressed in yeast is produced by Eurogentec SA in GMP conditions.

ELIGIBILITY:
All subjects had to meet the study inclusion criteria within 21 days prior to treatment,

Inclusion Criteria:

* Caucasian volunteers
* No smoker
* biological parameters (haematological, biochemical, renal and hepatic) in normal range
* Health Insurance
* sign inform consent

Exclusion Criteria:

* inflammatory or immunological pathology such as atopic diseases, evidence of inflammation or acute infection (including positive serology to viral hepatitis B and C or HIV)
* any immunological deficiency
* any clinically relevant alcohol or drug use (cannabis, opiates, cocaine, amphetamines, benzodiazepines, nicotine, barbiturates, meprobamate or antidepressant drugs according to urine drug and metabolites screen)
* current immunosuppressor treatment
* any other medication use within 2 weeks before the study
* any vaccination within the last 6 months
* no antibodies against Sh28GST protein.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1998-09; Primary Completion 1999-03 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D1 : administration, clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D21 : clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D28 : administration, clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D29 : clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D120 : clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D150 : administration, clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D165 : clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D180 : clinical observation, clinical analysis
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and rectal temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances

SECONDARY OUTCOMES:
Immunogenicity | Day of first administration and D21, D28, D29, D49, D120, D150, D165 and D180
  Immunogenicity was evaluated by dosage of specific antibody production, capacity of sera to inhibit enzymatic activity of the antigen, and immune profile estimation by in vitro cytokines production assay.

CONTACTS AND LOCATIONS:
Overall Officials: André CAPRON, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Gilles RIVEAU, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Christian LIBERSA, MD, Study Chair — CIC, University Hospital, Lille
Locations (1):
- Centre d'Investigation Clinique - CHRU de Lille, Lille, France

REFERENCES:
- [Background] Capron A, Riveau G, Capron M, Trottein F. Schistosomes: the road from host-parasite interactions to vaccines in clinical trials. Trends Parasitol. 2005 Mar;21(3):143-9. doi: 10.1016/j.pt.2005.01.003. PMID 15734662
- [Background] Capron A, Riveau GJ, Bartley PB, McManus DP. Prospects for a schistosome vaccine. Curr Drug Targets Immune Endocr Metabol Disord. 2002 Oct;2(3):281-90. doi: 10.2174/1568008023340587. PMID 12476492
- [Background] Capron A, Capron M, Riveau G. Vaccine development against schistosomiasis from concepts to clinical trials. Br Med Bull. 2002;62:139-48. doi: 10.1093/bmb/62.1.139. PMID 12176856
- [Result] Riveau G, Deplanque D, Remoue F, Schacht AM, Vodougnon H, Capron M, Thiry M, Martial J, Libersa C, Capron A. Safety and immunogenicity of rSh28GST antigen in humans: phase 1 randomized clinical study of a vaccine candidate against urinary schistosomiasis. PLoS Negl Trop Dis. 2012;6(7):e1704. doi: 10.1371/journal.pntd.0001704. Epub 2012 Jul 3. PMID 22802974